CLINICAL TRIAL: NCT01803477
Title: A Seamless Phase 1/2 Exploratory Multi-centre, Investigator-blind, Dose Escalation Study (Study Part 1), Followed by a Randomised, Intra-subject, Active Controlled Efficacy Study of Different Ingenol Mebutate Formulations Applied to the Forearm for 2 Consecutive Days (Study Part 2)
Brief Title: Safety and Dose Finding Study of New Vehicle Formulations Containing Ingenol Mebutate to Treat Actinic Keratosis on the Forearm
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LP0085-1000
Record Dates: First submitted 2013-02-28; First posted 2013-03-04 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2014-09

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate; Gels

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Picato® 0.05% gel (Active Comparator): once daily for two consecutive days
  Interventions: Drug: once daily for two consecutive days (Picato)
- ingenol mebutate vehicle formulation 1 (Experimental): once daily for two consecutive days
  Interventions: Drug: once daily for two consecutive days (Picato)
- ingenol mebutate vehicle formulation 2 (Experimental): once daily for two consecutive days
  Interventions: Drug: once daily for two consecutive days (Picato)
- ingenol mebutate vehicle formulation 3 (Experimental): once daily for two consecutive days
  Interventions: Drug: once daily for two consecutive days (Picato)

INTERVENTIONS:
Drug: once daily for two consecutive days (Picato)
  Other Names: Picato® 0.05% gel; escalating doses of ingenol mebutate vehicle formulation 1; escalating doses of ingenol mebutate vehicle formulation 2; escalating doses of ingenol mebutate vehicle formulation 3

SUMMARY:
The purpose of this study is to determine if the new vehicle formulations containing ingenol mebutate are as safe and effective as Picato® gel 0.05% (it's current vehicle formulation) when applied to AK lesions on the forearm for two consecutive days.

DETAILED DESCRIPTION:
This study will be run in 2 parts. The first part involves applying escalating concentrations of the new vehicle formulations containing ingenol mebutate to AKs on the forearms. Reactions and safety will be compared to Picato® (a registered and marketed ingenol mebutate gel) to ascertain if the new vehicle formulations are at least as safe and effective as Picato® . The purpose of part 2 is to select the concentration in the "new formulation" that produces this same, if not better response, as Picato® and with a similar or better safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Must be male or female and at least 18 years of age.
* Female patients must be of non-childbearing potential or if of childbearing potential then negative serum and urine pregnancy test and using effective contraception.
* Ability to provide informed consent.

Exclusion Criteria:

* location of the selected treatment area within 5cm of an incompletely healed wound or within 5cm of a suspected basal cell carcinoma or squamous cell carcinoma
* undergone Cosmetic or therapeutic procedures within 2cm of the selected treatment area in the 2 weeks prior to the treatment visit
* presence of sunburn within the selected treatment areas
* use of acid-containing therapeutic products within 2cm of the selected treatment area in the 2 weeks prior to the treatment visit
* previous enrolment in this clinical trial
* prior treatment with ingenol mebutate on the forearms
* use of topical moisturisers/creams/lotions, artificial tanners or topical steroids within 2cm of the selected treatment areas in the 2 weeks prior to the treatment visit
* treatment with immunomodulators, or interferon/interferon inducers or systemic medications that suppress the immune system within 4 weeks of the treatment visit
* treatment with 5-FU, imiquimod, diclofenac,or photodynamic therapy within 2 cm of the treatment area in the 8 weeks prior to the treatment visit
* use of systemic retinoids
* those who are currently participating in any other clinical trial
* females who are pregnant or are breastfeeding
* those known or suspected or not being able to comply with the requirements of the protocol or provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-02; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Safety of 3 new vehicle formulations containing ingenol mebutate compared to Picato® gel applied topically once daily for two consecutive days to four separate treatment areas containing actinic keratosis on the forearm | 2 weeks
  Safety data to be collected via CRF entries of AEs/SAEs and photographs. Relative skin reactions for comparison to Picato®.

SECONDARY OUTCOMES:
Evaluate treatment responses on AK of selected concentration of ingenol mebutate containing vehicle formulation from Part 1 compared to Picato® gel as assessed by reduction in the number of selected AK lesions 2 months after treatment | 2 months
  Assessed by visible and imaged lesion count

OTHER OUTCOMES:
Safety of the new ingenol mebutate vehicle formulation (ascertained in Part 1) compared to Picato® gel applied topically once daily for 2 consecutive days to 4 separate treatment areas containing actinic keratosis on the forearm | 8 weeks
  Safety data to be collected via CRF entries of AEs/SAEs and photographs. Treatment responses assessed by Reflective confocal microscopy scoring of visible selected AK lesions

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (2):
- Australia (2):
  - Dermatology Department, Woolloongabba, Queensland
  - Specialist Connect, Woolloongabba, Queensland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en
- See also: Therapeutic Goods Administration — http://www.tga.gov.au